CLINICAL TRIAL: NCT00676117
Title: A Single-Centre, Open, Randomised, Three-Way Cross-Over Drug-Drug Interaction Study of Esomeprazole (D961H) Capsule and Loxoprofen Tablet After Repeated Oral Administration in Japanese Healthy Male Subjects
Brief Title: Drug-Drug Interaction Study of Esomeprazole (D961H) Capsule and Loxoprofen Tablet After Repeated Oral Administration in Japanese Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind - Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D961HC00007
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: male; Japan; Japanese; Healthy volunteers
MeSH Terms: interventions — Esomeprazole; loxoprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Esomeprazole (D961H)
- 2 (Active Comparator)
  Interventions: Drug: Loxoprofen

INTERVENTIONS:
Drug: Esomeprazole (D961H) — 20mg
  Other Names: Nexium
  Arms: 1
Drug: Loxoprofen — 60mg tablet
  Other Names: Loxonin
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic profile of Esomeprazole (D961H) during repeated oral administration with and without co-administration of loxoprofen and the pharmacokinetic profile of loxoprofen during repeated oral administration with and without co-administration of Esomeprazole (D961H).

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male
* Body Mass Index (BMI=weight/height2) 19-27 (kg/m2)
* Body weight 50-80 kg

Exclusion Criteria:

* Past or present NSAIDs induced asthma, hepatic dysfunction, peptic ulcer or blood disorders
* Significant clinical illness from the 2 weeks preceding the pre-entry visit to the randomisation, as judged by the investigator(s) , eg, acute inflammatory disease which requires medical intervention
* Past or present cardiac, renal, hepatic, neurological or gastrointestinal disease, as judged by the investigator(s), eg, sequelae of myocardial infarction, nephritis, hepatitis and cerebral infarction

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic profile of D961H during repeated administration with and without co-administration of loxoprofen and pharmacokinetic profile of loxoprofen during repeated administration with and without co-administration of D961H, assessing plasma conc. | 5-7 days after the last dose of study medication is given

SECONDARY OUTCOMES:
The safety of D961H with and without coadministration of loxoprofen by assessment of adverse events, clinical laboratory tests (clinical chemistry, haematology, urinalysis and haemoccult test), ECG, blood pressure, pulse rate and body temperature | 5-7 days after the last dose of study medication is given

CONTACTS AND LOCATIONS:
Overall Officials: Naotsugu Oyama, MD, PhD, Study Director — AstraZeneca; Michio Yagi, Principal Investigator — Osaka Pharmacology Clinical Research Hospital
Locations (1):
- Research Site, Osaka, Osaka, Japan